CLINICAL TRIAL: NCT02105207
Title: Comparison Between Lung Ultrasound and Chest Radiography for Differential Diagnosis of Acute Dyspnea in the Emergency Department
Brief Title: Comparison Between Lung Ultrasound and Chest Radiography for Acute Dyspnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Enrico Lupia, MD, PhD, Assistant Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: iLUS-RCT
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Dyspnea; Congestive Heart Failure
MeSH Terms: conditions — Dyspnea; Heart Failure | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Ultrasound (Experimental): In Patients allocated to this arm Lung ultrasound for detection of interstitial syndrome will be performed before chest radiography.
  Interventions: Other: Lung Ultrasound
- Chest Radiography (Experimental): In Patients allocated to this arm chest radiography will be performed for the detection of indirect signs of pulmonary congestion/ADHF without ultrasound evaluation.
  Interventions: Other: Chest Radiography

INTERVENTIONS:
Other: Lung Ultrasound — Lung ultrasound evaluation is performed after clinical assessment and before chest radiography
  Arms: Lung Ultrasound
Other: Chest Radiography — Chest Radiography is performed after clinical evaluation without using ultrasound assessment
  Arms: Chest Radiography

SUMMARY:
For patients presenting to the Emergency Department with acute dyspnea, emergency physicians will be asked to categorize the diagnosis as acute decompensated heart failure or non-cardiogenic shortness of breath a) after the initial clinical assessment, and b) after performing lung ultrasound (LUS) for LUS arm or after chest radiography (CXR) and natriuretic peptide (NT-pro BNP) results for CXR arm. All patients will undergo CXR, those enrolled in the LUS arm, after sonographic evaluation. After discharge, the cause of patient's dyspnea will be determined by independent review of the entire medical records performed by two emergency physicians. In case of disagreement, a third expert physician will review entire medical records, and adjudicate the case.

DETAILED DESCRIPTION:
Study protocol After the initial standard work-up, which includes past medical history, history of the present illness, physical examination, ECG, and arterial blood gas analysis, the emergency physician responsible for patient care will be asked to categorize the diagnosis as ADHF or non-cardiogenic dyspnea.

Then, the patient will be assigned to one of the experimental arms. In the LUS arm, the same emergency physician will perform LUS, and express the new integrated presumptive etiology ("LUS-implemented" diagnosis). All patients will then undergo CXR.

In the CXR arm, patients will undergo CXR, and the new integrated etiology will be record after CXR and NT-proBNP results will be available.

After hospital discharge, two expert emergency physicians, blinded to LUS results, will independently review the entire medical record, and indicate the final diagnosis. In case of disagreement, a cardiologist will review the medical records, and adjudicate the case.

Statistical analysis The accuracy of each diagnostic tool will be expressed as sensitivity, specificity, predictive values and likelihood ratios obtained using 2 x 2 tables. "Positive" and "negative" results will be considered, for each test, the diagnosis of ADHF or non-cardiac dyspnea, respectively. Receiver operating characteristic (ROC) and area under curve (AUC) statistics will be also shown.

ELIGIBILITY:
Inclusion Criteria:

* acute dyspnea as chief complaint
* presence of an emergency physician skilled in lung ultrasound at evaluation time

Exclusion Criteria:

* mechanical ventilation ongoing at enrolment time
* dyspnea clearly related to a different aetiology (e.g. trauma, anxiety, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of Lung Ultrasound and Chest Radiography in dyspnoeic patients | Accuracy will be measured at the end of clinical evaluation in the Emergency Department, an expected average of 2 hours.
  Accuracy of lung ultrasound and chest radiography will be measured using as gold standard the independent evaluation of the entire medical records by two expert emergency physicians blinded to the lung ultrasound results and radiographic reports (digitalized chest radiography images will be available).

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Lupia, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (2):
- Italy (2):
  - Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - AOU Città della Salute e della Scienza di Torino, Turin

REFERENCES:
- [Background] Wang CS, FitzGerald JM, Schulzer M, Mak E, Ayas NT. Does this dyspneic patient in the emergency department have congestive heart failure? JAMA. 2005 Oct 19;294(15):1944-56. doi: 10.1001/jama.294.15.1944. PMID 16234501
- [Background] Niska R, Bhuiya F, Xu J. National Hospital Ambulatory Medical Care Survey: 2007 emergency department summary. Natl Health Stat Report. 2010 Aug 6;(26):1-31. PMID 20726217
- [Background] Peacock WF, Braunwald E, Abraham W, Albert N, Burnett J, Christenson R, Collins S, Diercks D, Fonarow G, Hollander J, Kellerman A, Gheorghiade M, Kirk D, Levy P, Maisel A, Massie BM, O'Connor C, Pang P, Shah M, Sopko G, Stevenson L, Storrow A, Teerlink J. National Heart, Lung, and Blood Institute working group on emergency department management of acute heart failure: research challenges and opportunities. J Am Coll Cardiol. 2010 Jul 27;56(5):343-51. doi: 10.1016/j.jacc.2010.03.051. PMID 20650354
- [Background] Ray P, Birolleau S, Lefort Y, Becquemin MH, Beigelman C, Isnard R, Teixeira A, Arthaud M, Riou B, Boddaert J. Acute respiratory failure in the elderly: etiology, emergency diagnosis and prognosis. Crit Care. 2006;10(3):R82. doi: 10.1186/cc4926. Epub 2006 May 24. PMID 16723034
- [Background] Redfield MM. Heart failure--an epidemic of uncertain proportions. N Engl J Med. 2002 Oct 31;347(18):1442-4. doi: 10.1056/NEJMe020115. No abstract available. PMID 12409548
- [Background] McCullough PA, Nowak RM, McCord J, Hollander JE, Herrmann HC, Steg PG, Duc P, Westheim A, Omland T, Knudsen CW, Storrow AB, Abraham WT, Lamba S, Wu AH, Perez A, Clopton P, Krishnaswamy P, Kazanegra R, Maisel AS. B-type natriuretic peptide and clinical judgment in emergency diagnosis of heart failure: analysis from Breathing Not Properly (BNP) Multinational Study. Circulation. 2002 Jul 23;106(4):416-22. doi: 10.1161/01.cir.0000025242.79963.4c. PMID 12135939
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Collins SP, Lindsell CJ, Storrow AB, Abraham WT; ADHERE Scientific Advisory Committee, Investigators and Study Group. Prevalence of negative chest radiography results in the emergency department patient with decompensated heart failure. Ann Emerg Med. 2006 Jan;47(1):13-8. doi: 10.1016/j.annemergmed.2005.04.003. Epub 2005 Jun 20. PMID 16387212
- [Background] Gillespie ND, McNeill G, Pringle T, Ogston S, Struthers AD, Pringle SD. Cross sectional study of contribution of clinical assessment and simple cardiac investigations to diagnosis of left ventricular systolic dysfunction in patients admitted with acute dyspnoea. BMJ. 1997 Mar 29;314(7085):936-40. doi: 10.1136/bmj.314.7085.936. PMID 9099117
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Liteplo AS, Marill KA, Villen T, Miller RM, Murray AF, Croft PE, Capp R, Noble VE. Emergency thoracic ultrasound in the differentiation of the etiology of shortness of breath (ETUDES): sonographic B-lines and N-terminal pro-brain-type natriuretic peptide in diagnosing congestive heart failure. Acad Emerg Med. 2009 Mar;16(3):201-10. doi: 10.1111/j.1553-2712.2008.00347.x. Epub 2009 Jan 29. PMID 19183402
- [Background] Picano E, Frassi F, Agricola E, Gligorova S, Gargani L, Mottola G. Ultrasound lung comets: a clinically useful sign of extravascular lung water. J Am Soc Echocardiogr. 2006 Mar;19(3):356-63. doi: 10.1016/j.echo.2005.05.019. PMID 16500505
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Noble VE, Murray AF, Capp R, Sylvia-Reardon MH, Steele DJR, Liteplo A. Ultrasound assessment for extravascular lung water in patients undergoing hemodialysis. Time course for resolution. Chest. 2009 Jun;135(6):1433-1439. doi: 10.1378/chest.08-1811. Epub 2009 Feb 2. PMID 19188552
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Background] Trovato GM, Sperandeo M. Sounds, ultrasounds, and artifacts: which clinical role for lung imaging? Am J Respir Crit Care Med. 2013 Apr 1;187(7):780-1. doi: 10.1164/ajrccm.187.7.780. No abstract available. PMID 23540884
- [Background] Anderson KL, Jenq KY, Fields JM, Panebianco NL, Dean AJ. Diagnosing heart failure among acutely dyspneic patients with cardiac, inferior vena cava, and lung ultrasonography. Am J Emerg Med. 2013 Aug;31(8):1208-14. doi: 10.1016/j.ajem.2013.05.007. Epub 2013 Jun 13. PMID 23769272
- [Background] Maisel A. B-type natriuretic peptide levels: diagnostic and prognostic in congestive heart failure: what's next? Circulation. 2002 May 21;105(20):2328-31. doi: 10.1161/01.cir.0000019121.91548.c2. No abstract available. PMID 12021215
- [Background] Januzzi JL, van Kimmenade R, Lainchbury J, Bayes-Genis A, Ordonez-Llanos J, Santalo-Bel M, Pinto YM, Richards M. NT-proBNP testing for diagnosis and short-term prognosis in acute destabilized heart failure: an international pooled analysis of 1256 patients: the International Collaborative of NT-proBNP Study. Eur Heart J. 2006 Feb;27(3):330-7. doi: 10.1093/eurheartj/ehi631. Epub 2005 Nov 17. PMID 16293638
- [Background] Cibinel GA, Casoli G, Elia F, Padoan M, Pivetta E, Lupia E, Goffi A. Diagnostic accuracy and reproducibility of pleural and lung ultrasound in discriminating cardiogenic causes of acute dyspnea in the emergency department. Intern Emerg Med. 2012 Feb;7(1):65-70. doi: 10.1007/s11739-011-0709-1. Epub 2011 Oct 28. PMID 22033792
- [Background] Knudsen CW, Omland T, Clopton P, Westheim A, Abraham WT, Storrow AB, McCord J, Nowak RM, Aumont MC, Duc P, Hollander JE, Wu AH, McCullough PA, Maisel AS. Diagnostic value of B-Type natriuretic peptide and chest radiographic findings in patients with acute dyspnea. Am J Med. 2004 Mar 15;116(6):363-8. doi: 10.1016/j.amjmed.2003.10.028. PMID 15006584
- [Background] Gargani L, Frassi F, Soldati G, Tesorio P, Gheorghiade M, Picano E. Ultrasound lung comets for the differential diagnosis of acute cardiogenic dyspnoea: a comparison with natriuretic peptides. Eur J Heart Fail. 2008 Jan;10(1):70-7. doi: 10.1016/j.ejheart.2007.10.009. PMID 18077210
- [Background] Garcia X, Simon P, Guyette FX, Ramani R, Alvarez R, Quintero J, Pinsky MR. Noninvasive assessment of acute dyspnea in the ED. Chest. 2013 Aug;144(2):610-615. doi: 10.1378/chest.12-1676. PMID 23471509
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404
- [Background] Eurlings LW, Sanders-van Wijk S, van Kimmenade R, Osinski A, van Helmond L, Vallinga M, Crijns HJ, van Dieijen-Visser MP, Brunner-La Rocca HP, Pinto YM. Multimarker strategy for short-term risk assessment in patients with dyspnea in the emergency department: the MARKED (Multi mARKer Emergency Dyspnea)-risk score. J Am Coll Cardiol. 2012 Oct 23;60(17):1668-77. doi: 10.1016/j.jacc.2012.06.040. Epub 2012 Sep 26. PMID 23021334